CLINICAL TRIAL: NCT03538197
Title: SURAYA : Suicide Re Attempts in Young Adults After First Suicide Attempt : Socio-demographic, Clinical and Biological Correlates
Brief Title: Suicide Re Attempts in Young Adults After First Suicide Attempt : Socio-demographic, Clinical and Biological Correlates
Acronym: SURAYA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hôpital le Vinatier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2017-A03129-44
Record Dates: First submitted 2018-04-16; First posted 2018-05-29 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Suicide
Keywords: suicide attempt; suicide re attempt
MeSH Terms: conditions — Suicide; Suicide, Attempted

STUDY DESIGN:
Intervention Model Description: Cohort study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SUICID ATTEMPT YOUNG PEOPLE (Other): Suicide Re Attempts in Young Adults after first suicide attempt : socio-demographic, clinical and biological correlates
  Interventions: Other: clinical and biological correlates

INTERVENTIONS:
Other: clinical and biological correlates — To measure the rate of suicidal re attempt (SR) in a population of young adults aged 18 to 25 years.
  To identify sociodemographic, clinical and biological characteristics of a population of suicidal young people, in an attempt to highlight potential risk factors

SUMMARY:
Suicide is the second leading cause of death among people aged 15 to 24 (WHO, 2014). After a first suicide attempt, the 18 to 25 years old would be very likely to repeat the act: 25 to 31% would make a new attempt in the following year (Christiansen et al, 2007).

Nevertheless the literature on this subject is not detailed. In this project, we hypothesize that young adults aged 18 to 25 who have made their first suicide attempt will repeat their act more frequently than younger or older populations. In addition, these young people would have identifiable risk factors (sociodemographic, clinical and biological) that differ from young people who do not enter this phenomenon.

Our main objective is to measure the rate of suicidal reiteration in a population of young adults aged 18 to 25 years.

Our secondary objectives are to identify sociodemographic, clinical and biological characteristics of a population of suicidal re attempt young people, to highlight potential risk factors

DETAILED DESCRIPTION:
Objectives:

* Our main objective is to measure the rate of suicidal re attempt (SR) in a population of young adults aged 18 to 25 years.
* Our secondary objectives are to identify sociodemographic, clinical and biological characteristics of a population of suicidal young people, in an attempt to highlight potential risk factors. We will try to highlight correlations between the reiteration of the suicidal act and:

  1. socio-demographic criteria: level of urbanity, socio-economic level, social and family context, date and place of birth, religion, sexual orientation, name and contact details of the general practitioner, previous access to care
  2. scores on the scales of various psychiatric pathologies, existing or in formation (eg depression, anxiety disorders, psychosis)
  3. alterations at the peripheral level
* on the stress response system: cortisolemia and capillary cortisol levels
* on the total and mature serum BDNF

In addition, DNA and RNA genetic samples will be taken in order to constitute a biological collection for later research.

Type of study: This is an interventional research with minimal risks and constraints (2 ° study), multicenter prospective cohort.

Number of centers: 2 Suicide Prevention Center at the Le Vinatier Hospital Center and the Post Crisis Unit at the Edouard Herriot Hospital of the Hospices Civils de Lyon.

Description of the study / experimental plan:

This is a prospective cohort study that will be divided into two groups: "repeat suicide attempt" and "no repeat attempt"

Primary judgment criterion:

This is the occurrence of repeating a suicide attempt (over a period of 3 months after the initial attempt.

In this project, a suicide attempt is defined according to WHO criteria as "non-fatal suicidal behavior, self-inflicted injury with a desire to end one's life that does not lead to death".

Number of subjects:

Our study will include 200 patients at the Le Vinatier CH Suicide Prevention Center and the Post Crisis Unit at Edouard Herriot Hospital.

inclusion criteria: between the ages of 18 and 25

* a first suicide attempt
* Master French sufficient

Exclusion Criteria:

-Majors protected: under curatorship or under guardianship

Course of the study :

-Inclusion will take place immediately after the first suicide attempt at the Post Crisis Unit at Edouard Herriot Hospital and the Suicide Prevention Center.

An anamnestic collection of social and demographic data will be carried out: level of urbanity, professional activity, level of study, access to care, and previous care received, socio-economic level, social and family context (notably existing conflict with parents or love break-up). The patient's telephone number will be collected as well as the patient's psychiatric and addiction history, and the means used for the suicide attempt.

Different scales of assessments, by means of self-questionnaires, will be given to the patient and an investigator will provide the C-SSRS scale assessment for the suicidal risk severity. Finally a venous blood sample will be performed with a measure of total and mature serum BDNF and cortisolemia. Capillary cortisol will also be measured.

After obtaining the patient's consent, two blood samples (DNA and RNA) will be collected and stored at -80 degrees to create a biological collection for later research.

An orientation in the course of care will then be given to the subject who will receive the appropriate care as well as a phone call made by the Suicide Prevention Center.

-At 3 months: A phone call will be made to check the presence or absence of the main evaluation criterion: the repetition of a suicide attempt. In addition, the patient will be asked about life events during these three months and the care received since inclusion.

Benefits and risks of this study:

The expected benefits of this study are: a better understanding of the mechanisms underlying the recurrence of the suicidal act, which could allow an optimal patient management and an adapted orientation in the care network, this for a setting in place in the near future.

In addition, patients included in the study will benefit from follow-up.

The foreseeable risk is the SR that can lead to suicide. To minimize this risk, each patient included in this protocol will benefit from a clinical evaluation performed by a trained investigator. At the end of this evaluation, according to the observed suicidal risk, an orientation in the course of care will be proposed. Each patient will be informed of the different modalities of psychiatry consultations and how to challenge the network. In addition, all patients will receive a phone call from the Suicide Prevention Center.

No serious adverse effects that could be attributed to the project are expected as part of this research.

Indeed, the blood test is carried out systematically as part of a post-suicide treatment and no other invasive examination is scheduled. The only undesirable events that can occur after a venous blood collection are: a hematoma at the point of puncture, pain during the bite, vagal discomfort or rare cases of infectious risks. These risks are greatly minimized by means of sterile single-use equipment and qualified medical personnel, and can not be considered as a serious expected adverse effect.

ELIGIBILITY:
Inclusion Criteria:

* between the ages of 18 and 25
* a first suicide attempt
* Master French sufficient

Exclusion Criteria:

* Majors protected: under curatorship or under guardianship

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2018-05-22 (Actual); Primary Completion 2022-06-29 (Actual); Study Completion 2022-06-29 (Actual)

PRIMARY OUTCOMES:
Assessment of the prevalence of SR rate over a 3-months period after the first suicide attempt, among young adults aged 18 to 25. | Within the first 3 months following a first suicide attempt

SECONDARY OUTCOMES:
mature and total BDNF | Within the first 3 months after the first suicide attempt
  We will try to highlight correlations between the reiteration of the suicidal act and biological measures
level of urbanity | Within the first 3 month following a first suicide attempt
  sociodemographic risk factor
socio-economic level | Within the first 3 month following a first suicide attempt
  sociodemographic risk factor
social and family context | Within the first 3 months following a first suicide attempt
  sociodemographic risk factor
date of birth | Within the first 3 months following a first suicide attempt
  sociodemographic risk factor
place of birth | Within the first 3 months following a first suicide attempt
  sociodemographic risk factor
BIS : Barratt Impulsive Scale | Within the first 3 months following a first suicide attempt
  The Barratt Impulsiveness Scale (BIS) is a widely used measure of impulsiveness. It includes 30 items that are scored to yield six first-order factors (attention, motor, self-control, cognitive complexity, perseverance, and cognitive instability impulsiveness) and three second-order factors (attentional, motor, and non-planning impulsiveness).
  Clinical risk factor : We aim to highlight correlations between the reiteration of the suicidal act and different scores on clinical scales
C-SSRS : Colombia Suicide Severity Rating Scale | Within the first 3 months following a first suicide attempt
  The Screener contains 6 "yes" or "no" questions in which respondents are asked to indicate whether they have experienced several thoughts or feelings relating to suicide over the past month and behaviors over their lifetime and past 3 months. Each question addresses a different component of the respondent's suicide ideation severity and behavior.
  Question 1: wish to be dead Question 2: non-specific suicidal thoughts Questions 3-5: more specific suicidal thoughts and intent to act Question 6: suicidal behavior over the respondent's lifetime and past 3 months If the respondent answers "yes" to Question 2, he/she is instructed to answer Questions 3-5. If the respondent answers "no" to Question 2, he/she may skip to Question 6.
  An answer of "yes" to any of the six questions may indicate a need for referral to a trained mental health professional and an answer of "yes" to questions 4, 5 or 6 indicate high-risk.
hair cortisol and blood cortisol | Within the first 3 months following a first suicide attempt
  We will try to highlight correlations between the reiteration of the suicidal act and biological measures
Analog visual scales | Within the first 3 months following a first suicide attempt
  The visual analogue scale or visual analog scale (VAS) is a psychometric response scale which can be used in questionnaires. It is a measurement instrument for subjective characteristics or attitudes that cannot be directly measured. When responding to a VAS item, respondents specify their level of agreement to a statement by indicating a position along a continuous line between two end-points.
  Clinical risk factor : We aim to highlight correlations between the reiteration of the suicidal act and different scores on clinical scales
Negative life events during the last 6 months | Within the first 3 months following a first suicide attempt
  Clinical risk factor : We aim to highlight correlations between the reiteration of the suicidal act and different scores on clinical scales
The reasons for living inventory | Within the first 3 months following a first suicide attempt
  Clinical risk factor : We aim to highlight correlations between the reiteration of the suicidal act and different scores on clinical scales
CTQ : childhood trauma questionnary | Within the first 3 months following a first suicide attempt
  Clinical risk factor : We aim to highlight correlations between the reiteration of the suicidal act and different scores on clinical scales
STAXI-2 | Within the first 3 months following a first suicide attempt
  Clinical risk factor : We aim to highlight correlations between the reiteration of the suicidal act and different scores on clinical scales
PQB : psychosis risk screening | Within the first 3 months following a first suicide attempt
  Clinical risk factor : We aim to highlight correlations between the reiteration of the suicidal act and different scores on clinical scales
QIDS : Quick Inventory of Depressive Symptomatology | Within the first 3 months following a first suicide attempt
  Clinical risk factor : We aim to highlight correlations between the reiteration of the suicidal act and different scores on clinical scales
MDQ : Mood disorder questionnaire | Within the first 3 months following a first suicide attempt
  Clinical risk factor : We aim to highlight correlations between the reiteration of the suicidal act and different scores on clinical scales
CUDIT : Cannabis use Disorders Identification Test | Within the first 3 months following a first suicide attempt
  Clinical risk factor : We aim to highlight correlations between the reiteration of the suicidal act and different scores on clinical scales
CAST : Cannabis Abuse Screening Test | Within the first 3 months following a first suicide attempt
  Clinical risk factor : We aim to highlight correlations between the reiteration of the suicidal act and different scores on clinical scales
Fagerstrom Questionary | Within the first 3 months following a first suicide attempt
  Clinical risk factor : We aim to highlight correlations between the reiteration of the suicidal act and different scores on clinical scales
AUDIT : Alcohol use disorders test | Within the first 3 months following a first suicide attempt
  Clinical risk factor : We aim to highlight correlations between the reiteration of the suicidal act and different scores on clinical scales

CONTACTS AND LOCATIONS:
Overall Officials: POULET Emmanuel, Ph, Principal Investigator — CH LE VINATIER
Locations (1):
- Centre Hospitalier Le Vinatier, Bron, AURA, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Abrial E, Chalancon B, Leaune E, Brunelin J, Wallon M, Moll F, Barakat N, Hoestlandt B, Fourier A, Simon L, Magnin C, Hermand M, Poulet E. Investigating Predictive Factors of Suicidal Re-attempts in Adolescents and Young Adults After a First Suicide Attempt, a Prospective Cohort Study. Study Protocol of the SURAYA Project. Front Psychiatry. 2022 Jun 29;13:916640. doi: 10.3389/fpsyt.2022.916640. eCollection 2022. PMID 35845461